CLINICAL TRIAL: NCT05764629
Title: An Observational Study of Risk Factors Influencing Glycemic Status and Optimized Treatment on Post-chronic Pancreatitis Diabetes Mellitus
Brief Title: An Observational Study on Post-chronic Pancreatitis Diabetes Mellitus
Status: Active, not recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Principal Investigator, Changhai Hospital
Other Study IDs: PPDM-C
Record Dates: First submitted 2023-02-18; First posted 2023-03-10 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pancreatitis; Diabetes Mellitus
MeSH Terms: conditions — Pancreatitis, Chronic; Diabetes Mellitus | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The peripheral blood sample for laboratory examinations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood test — Testing the peripheral blood for PPDM-C, including blood glucose, glycated hemoglobin A1c, fasting insulin and C-peptide, etc.
Drug: pharmacologic approaches to glycemic treatment — documenting the change of glycemic treatment during the follow-up period

SUMMARY:
To explore the risk factors influencing glycemic status, optimized treatment, and prognosis of post-chronic pancreatitis diabetes mellitus (PPDM-C).

DETAILED DESCRIPTION:
The present study was an observational study aimed to explore risk factors influencing glycemic status, optimized treatment, and prognosis of post-chronic pancreatitis diabetes mellitus. The observation items included clinical characteristics, blood glucose control and incidence of complications of PPDM-C.

ELIGIBILITY:
Inclusion Criteria:

1. patients with diagnosis of chronic pancreatitis and diabetes mellitus.
2. participants with painless chronic pancreatitis were diagnosed with diabetes within 2 years of the diagnosis of chronic pancreatitis.
3. participants with painful chronic pancreatitis were diagnosed with diabetes after the first attack of chronic pancreatitis.

Exclusion Criteria:

1. participants with suspected malignant tumors of the pancreas or other sites of body, or participants in the terminal stage of severe disease
2. serious mental illness, lesion of liver or kidney, pregnancy, breast-feeding or planning pregnancy
3. definitely diagnosed type 1 diabetes, type 2 diabetes, or other metabolic diseases that affect blood glucose
4. autoimmune pancreatitis
5. Scarcity of information related to HbA1c
6. death or loss of follow-up during follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consequent patients with a diagnosis of PPDM-C in Changhai Hospital between 2018 to 2022
Sampling Method: Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) | through study completion, an average of 1 year
  measure the control of blood glucose of every 3 months

SECONDARY OUTCOMES:
Adverse events | through study completion, an average of 1 year
  Incidence and frequency (number of events) of adverse events (%) such as hypoglycemia, cardiovascular disease, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided